CLINICAL TRIAL: NCT07230418
Title: A Double-blind, Randomized, Dose-escalation Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of Single and Multiple Doses of HRS-3095 Oral Administration in Healthy Subjects, as Well as the Effect of HRS-3095 on CYP3A4 Metabolic Enzymes
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of Single and Multiple Doses of HRS-3095 Oral Administration in Healthy Subjects, as Well as the Effect of HRS-3095 on CYP3A4 Metabolic Enzymes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-3095-101
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-3095 Group (Experimental)
  Interventions: Drug: HRS-3095 Tablet
- HRS-3095 Placebo Group (Placebo Comparator)
  Interventions: Drug: HRS-3095 Placebo Tablet

INTERVENTIONS:
Drug: HRS-3095 Tablet — Oral HRS-3095 tablet.
  Arms: HRS-3095 Group
Drug: HRS-3095 Placebo Tablet — Oral HRS-3095 placebo tablet.
  Arms: HRS-3095 Placebo Group

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple doses of HRS-3095 oral administration in healthy subjects. This study will also explore food effect and the effect of HRS-3095 on CYP3A4 metabolic enzymes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form (ICF);
2. Male and female healthy subjects with an age range between 18 and 55 years (inclusive);
3. Body mass index between 18.0 and 32.0 kg/m2 (inclusive), and the body weight is ≥ 50 kg for men and ≥ 45 kg for women;
4. For healthy subjects, no clinically significant abnormalities;
5. Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods.

Exclusion Criteria:

1. Known medical history or clinical manifestation of circulatory, endocrine, neurological, digestive, respiratory, hematological, immunological, psychiatric diseases, metabolic disorders, or any other condition that may interfere with the trial results, as determined by the Investigator;
2. Any condition or disease that may affect drug absorption, distribution, metabolism, or excretion, as determined by the Investigator;
3. History of recurrent drug allergies, or a physician-diagnosed and treatment-requiring allergic disease, or known allergy to any component of the investigational product;
4. History of an infection requiring systemic antimicrobial therapy within 2 weeks prior to screening or within 2 weeks before the first dose of the investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 21 days.
Incidence of serious adverse events (SAEs) | Up to 21 days.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Up to 17 days.
Time of maximum concentration (Tmax) | Up to 17 days.
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) | Up to 17 days.
Area under the concentration-time curve from time zero to infinity (AUC0-inf) | Up to 17 days.
Area under the concentration-time curve from time zero to the end of the dosing interval tau (AUC0-tau) | Up to 17 days.
Elimination half-life (t1/2) | Up to 17 days.
Apparent clearance (CL/F) | Up to 17 days.
Apparent volume of distribution (Vz/F) | Up to 17 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Frist Clinical Medicial College of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided